CLINICAL TRIAL: NCT01544244
Title: Comparison of the Global Shoulder Concept (GSC) Method Versus Classic Physical Therapy for Shoulder Tendinitis: a Prospective, Randomized Study
Brief Title: The Global Shoulder Concept (GSC) Method Versus Classic Physical Therapy for Shoulder Tendinitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion curve too slow.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRIP/2011/DR-03; 2011-A01168-33 (Other: RCB number)
Record Dates: First submitted 2012-02-23; First posted 2012-03-05 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Shoulder; Tendinopathy
Keywords: comparison of physical therapy strategies
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSC physcial therapy (Experimental): Patients included in this arm of the study will follow the Global Shoulder Concept physical therapy sequence.
  Interventions: Procedure: GSC physical therapy
- Standard (Active Comparator): Patients in this arm of the study will follow the standard physical therapy sequence.
  Interventions: Procedure: Standard physical therapy

INTERVENTIONS:
Procedure: GSC physical therapy — Global Shoulder Concept physical therapy sequence for shoulder tendonitis. The procedures used in this protocol refer to physical therapy sequences, not to devices or drugs.
  Arms: GSC physcial therapy
Procedure: Standard physical therapy — Standard physical therapy sequence for shoulder tendonitis. The procedures used in this protocol refer to physical therapy sequences, not to devices or drugs.
  Arms: Standard

SUMMARY:
The primary objective of this study is to demonstrate the superiority of the CGE physical therapy protocol versus a standard physical therapy protocol of the shoulder by measuring the following after 1 month of physical therapy: the FI2S score including validated measures of pain, glenohumeral joint range of motion in the three planes, the ability to perform certain everyday activities and the strength of forward elevation measured with a dynamometer.

DETAILED DESCRIPTION:
Secondary objectives:

* To study the evolution of passive glenohumeral range of motion
* To study the evolution of the global range of passive and active motion for each method used
* To evaluate functional recovery (DASH)
* To evaluate the impact on quality of life (SF36)
* To study the difference in visual analog scale scores for pain during physical therapy sessions
* Compare the two methods/groups after three months.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* painful, chronic tendinopathy (more than 3 months) of the rotator cuff, confirmed by MRI

Exclusion Criteria:

* The patient is pregnant or breastfeeding
* Any emergency situation
* Non-mechanical tendinopathies (metabolic, neurological, capsulitis, reflex sympathetic dystrophy) and tendon surgery (tendon surgery and acromioplasty)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
change in FI2S score | 90 days

SECONDARY OUTCOMES:
Change in visual analog scale for pain | Day 1 versus baseline
Change in visual analog scale for pain | Day 5 versus baseline
Change in visual analog scale for pain | Day 12 versus baseline
Change in visual analog scale for pain | Day 19 versus baseline
Change in visual analog scale for pain | Day 26 versus baseline
Change in visual analog scale for pain | Day 90 versus baseline
Scapulohumeral amplitude gain in 3 main directions | Day 1
  Passive and active mobility are evaluated by manual goniometry.
Scapulohumeral amplitude gain in 3 main directions | Day 26
  Passive and active mobility are evaluated by manual goniometry.
Scapulohumeral amplitude gain in 3 main directions | Day 90
  Passive and active mobility are evaluated by manual goniometry.
Functional gain as measured by the DASH self questionnaire | Day 1
Functional gain as measured by the DASH self questionnaire | Day 5
Functional gain as measured by the DASH self questionnaire | Day 12
Functional gain as measured by the DASH self questionnaire | Day 19
Functional gain as measured by the DASH self questionnaire | Day 26
Functional gain as measured by the DASH self questionnaire | Day 90
FI2S score | Day 1
FI2S score | Day 5
FI2S score | Day 12
FI2S score | Day 19
FI2S score | Day 26
SF36 self questionnaire | Day 1
SF36 self questionnaire | Day 26
SF36 self questionnaire | Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Richard, Study Director — Centre Hospitalier Universitaire de Nîmes; Arnaud Dupeyron, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes